CLINICAL TRIAL: NCT07370480
Title: Evaluation of the Effectiveness of the Enghien-les-Bains Thermal Spa Treatment in the Rheumatology Indication in Patients With Knee Osteoarthritis. Indirect Comparison Study.
Brief Title: Knee Osteoarthritis and Thermal Spa Treatment
Acronym: ENERGIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: Town Hall of Enghien-les-Bains (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1757; 2025-A00448-41 (Other: French Competent Authority (ANSM))
Record Dates: First submitted 2026-01-13; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: spa therapy; thermal treatment; balneotherapy; Rheumatology
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Water Pollution; Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, superiority study with external comparison (control group of a reference RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal spa treatment (Experimental): 18-day spa program with Waters of Enghien-les-Bains in addition to standard of care for knee osteoarthritis
  Interventions: Other: Thermal spa sessions; Other: Thermal water; Other: Standard of Care for Knee Osteoarthritis

INTERVENTIONS:
Other: Thermal spa sessions — At least 4 spa sessions per day, 6 days a week during 3 consecutive weeks that may include daily: one whirlpool bath, one poultice application, one overall jet shower and one underwater massage with thermal water.
  With the exception of the application of mud poultices and whirlpool bath, which cannot be substituted, other treatments may be replaced by: immersion bath with shower, penetrating shower, and local jet shower.
  10-minute air diffusion baths are taken in individual tubs at 37°C. Mud is applied for 10 minutes as a poultice to both knees (minimum 2 per knee, 45°C), if necessary, to other painful osteoarthritis areas. A 3-minute overall jet shower is administered by a thermal spa staff member, using thermal water at 37°C. A 10-minute underwater massage is administered by a physiotherapist, under a thermal water spray bar at 37°C.
Other: Thermal water — The water has a neutral pH (7), is cold (14 °C), and presents a moderate level of mineralization (571 mg/L) with a balanced ionic profile. It contains calcium (128 mg/L), bicarbonates (440 mg/L), sulfates (93 mg/L), magnesium (27.9 mg/L), and sodium (12.4 mg/L).
  Other Names: Natural Mineral Water of Enghiens-les-Bains
Other: Standard of Care for Knee Osteoarthritis — Participants continue standard medical care for knee osteoarthritis as prescribed by their primary care physician, including analgesics and physiotherapy, according to routine clinical practice.

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness at 6 months of the Enghien-les-Bains thermal spa treatment on functional disability and pain, assessed by the Minimal Clinically Important Improvement (MCII), in patients with knee osteoarthritis.

The study is conducted in patients aged 50 to 80 years with knee osteoarthritis (Kellgren-Lawrence grade 2 to 4) and a baseline functional impairment defined by a normalized WOMAC function score ≥ 30.

The main questions it aims to answer are:

* Does the Enghien-les-Bains thermal spa treatment result in a clinically meaningful improvement in pain and functional disability at 6 months in patients with knee osteoarthritis?
* Is the effectiveness of the Enghien-les-Bains thermal spa treatment superior to standard care, as assessed through an indirect comparison with an external control group from the ANGELLO randomized controlled trial (NCT0581943)? Patients receiving the Enghien-les-Bains thermal spa treatment are compared to the external control group of the ANGELLO randomized controlled trial (Saint-Jean-d'Angély), composed of non-spa-treated patients receiving standard care, to assess differences in pain and functional disability outcomes at 6 months.

Patients of the study:

* Undergo a standardized thermal spa treatment at Enghien-les-Bains.
* Continue usual medical care for knee osteoarthritis.
* Complete questionnaires and clinical assessments at baseline and at 6 months.

DETAILED DESCRIPTION:
This study includes three medical visits with the investigator: one within 28 days before the thermal spa treatment, one at the end of the treatment, and one 6 months after the start of the treatment. At inclusion, informed consent is obtained, eligibility criteria are verified, and baseline data are collected, including self-administered questionnaires assessing pain, function, and quality of life before the start of the treatment.

During the 20-day thermal spa treatment, care provided and any adverse events are recorded. Clinical assessments and questionnaires are repeated at the end of the treatment. Additional patient-reported outcomes and treatment changes are collected at 3 months, and a final clinical evaluation and questionnaires are completed at 6 months.

An ancillary qualitative study evaluates the conditions under which the thermal spa treatment program is effective from the participants' perspective, including their engagement, lived experience, perceived benefits, facilitators and barriers, and any adaptations made. Data are collected through individual semi-structured face-to-face interviews at the end of the treatment, which are audio-recorded, fully transcribed, and qualitatively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis with Kellgren and Lawrence stage 2 to 4 evidenced by a knee X-ray examination in the past 3 years.
* 100-normalized score of the WOMAC physical function subscale greater than or equal to 30.
* Signed inform consent.
* With health insurance affiliation.

Exclusion Criteria:

* Presented with balneotherapy contraindication or to certain adjuvant treatment techniques (balneation, hydrotherapy jets, massage): chronic infectious pathology, active cancer, decompensated cardiac, hepatic or renal insufficiency, "open" leg ulcer, immune deficiency, phlebitis, erysipelas or history of erysipelas, active thrombosis, behavioral disorders, etc.
* Presented with chronic pain for reasons other than osteoarthritis: chronic inflammatory rheumatism (rheumatoid arthritis, ankylosing spondylitis, lupus, psoriatic arthritis) or fibromyalgia.
* Patient scheduled for knee osteoarthrosis-related surgery within the next 7 months.
* Having had spa treatment in the past 6 months whatever the indication or intra-articular corticosteroid injection within the previous 90 days or hyaluronic acid infiltration or other viscosupplementation or platelet-rich plasma (PRP) injection within the previous 6 months.
* Having planned a spa treatment in another indication between inclusion and final visit.
* Residing more than 30 kilometers from Enghien-les-Bains at the time of spa treatment.
* Women of childbearing potential who are not using effective contraception (estrogen/progestin or progestin-only oral, vaginal, transdermal, injectable or subcutaneous) or who plan to discontinue contraception within the next 7 months.
* Likely to be unable to comply with protocol or to attend visits, particularly in view of the duration of the research, or unable to read or understand French.
* Regulatory reason (guardianship or already enrolled in a clinical trial).
* Already included in a clinical trial or in the exclusion period of a clinical trial.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Clinically Important Improvement (MCII) at 6 months | 6 months
  MCII is defined as a pain reduction of 19.9 mm or more on a 0-100 visual analogic scale (VAS), where 0 means no pain and 100 worse pain.
  The percentage of patients achieving MCII is calculated and compared with that of the control group in the reference RCT (external comparison).
Minimal Clinically Important Improvement (MCII) at 6 months | 6 months
  MCII is defined as a reduction of 9.1 points or more in the function subscale of the Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) in absence of knee surgery. WOMAC is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations).
  The percentage of patients achieving MCII is calculated and compared with that of the control group in the reference RCT (external comparison).

SECONDARY OUTCOMES:
Change from baseline of pain-related knee osteoarthritis at 20 days | Day 1 and 20 days
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of pain-related knee osteoarthritis at 3 months | Day 1 and 3 months
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of pain-related knee osteoarthritis at 6 months | Day 1 and 6 months
  Pain intensity is measured using a 0 (no pain)-100 (Worse pain) Visual Analogic Scale (VAS). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of the pain subscale of the WOMAC at 20 days | Day 1 and 20 days
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of the pain subscale of the WOMAC at 3 months | Day 1 and 3 months
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of the pain subscale of the WOMAC at 6 months | Day 1 and 6 months
  Pain subscale of the WOMAC is a self-administered questionnaire that consists in 5 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse pain limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of stiffness subscale of the WOMAC at 20 days | Day 1 and 20 days
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of stiffness subscale of the WOMAC at 3 months | Day 1 and 3 months
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of stiffness subscale of the WOMAC at 6 months | Day 1 and 6 months
  Stiffness subscale of the WOMAC is a self-administered questionnaire that consists in 2 items: during walking, using stairs, in bed, sitting or lying, and standing upright. The 100-normalized subscale score ranges from 0 (none) to 100 (worse stiffness limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of physical function subscale of the WOMAC at 20 days | Day 1 and 20 days
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of physical function subscale of the WOMAC at 3 months | Day 1 and 3 months
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of physical function subscale of the WOMAC at 36 months | Day 1 and 6 months
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of physical function subscale of the WOMAC at 6 months | Day 1 and 6 months
  Physical function subscale of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire that consists in 17 items: (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. The 100-normalized subscale score ranges from 0 (none) to 100 (worse functional limitations). Mean variation is compared with that of the control group in the reference RCT (external comparison).
Change from baseline of total score of the WOMAC at 20 days | Day 1 and 20 days
  The scores for each of the 3 subscales (function, pain, stiffness) are summed up to calculate the total WOMAC score. The 100-normalized score ranges from 0 (none) to 100 (worse limitations).
Change from baseline of total score of the WOMAC at 6 months | Day 1 and 6 months
  The scores for each of the 3 subscales (function, pain, stiffness) are summed up to calculate the total WOMAC score. The 100-normalized score ranges from 0 (none) to 100 (worse limitations).
Changes from baseline of quality of life at 20 days | Day 1 and 20 days
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes patient health state. Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of quality of life at 3 months | Day 1 and 3 months
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes patient health state. Mean variation is compared with that of the control group in the reference RCT (external comparison).
Changes from baseline of quality of life at 6 months | Day 1 and 6 months
  Quality of life is measured using EUROQOL (EQ-5D-3L) questionnaire. The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes patient health state. Mean variation is compared with that of the control group in the reference RCT (external comparison).
Acceptable Symptom State (ASS) at 20 days | Day 20
  ASS is defined as VAS pain value of 32 mm or less or a WOMAC function subscale, normalized to a 0-100 score of 31 points or less. The percentage of patients achieving ASS is calculated and compared with that of the control group in the reference RCT (external comparison).
Acceptable Symptom State (ASS) at 3 months | 3 months
  ASS is defined as VAS pain value of 32 mm or less or a WOMAC function subscale, normalized to a 0-100 score of 31 points or less. The percentage of patients achieving ASS is calculated and compared with that of the control group in the reference RCT (external comparison).
Acceptable Symptom State (ASS) at 6 months | 6 months
  ASS is defined as VAS pain value of 32 mm or less or a WOMAC function subscale, normalized to a 0-100 score of 31 points or less. The percentage of patients achieving ASS is calculated and compared with that of the control group in the reference RCT (external comparison).
Management of knee osteoarthritis over the study | 6 months
  Number and frequency of treatments for knee osteoarthritis (analgesics, chondro-protectors or antarthritics, intra-articular injections of corticoids and hyaluronic acid, physical or surgical treatments). Numbers and frequencies of treatments are compared with those of the control group in the reference RCT (external comparison).
Safety of the18-day spa treatment (therapeutic indication: Rheumatology) at Enghien-les-Bains | 6 months
  Adverse effects related to the spa treatment are described using MedDRA, whether they occurred during or after the 18-day spa treatment.

OTHER OUTCOMES:
Qualitative assessment of participant experience and engagement with the thermal spa treatment | Day 20
  Semi-structured individual interviews are conducted with a subset of participants to explore their level of engagement, lived experience, and perceived benefits of the thermal spa treatment. The interviews also assess facilitators and barriers encountered during participation, as well as any adaptations made by participants, from their own perspective. Interview data are analyzed using qualitative thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Magali Ballard, MD, Principal Investigator
Locations (2):
- France (2):
  - Thermes d'Enghien-les-Bains, Enghien-les-Bains
  - Thermes d'Enghien-les-Bains, Enghien-les-Bains, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No
The informed consent obtained from participants does not include provisions for sharing individual participant data with external researchers.

REFERENCES:
- [Background] Grant L. Oil, Egypt and Israel: the view in 1995. NPG Forum Ser. 1991 Apr:1-4. PMID 12178974